CLINICAL TRIAL: NCT04326556
Title: Individual and Environmental Risk Factors for Unscheduled Hospitalizations of Elderly People, With Sensor-based Measurements of the Peri-individual Environment: a Prospective Cohort
Brief Title: Individual and Environmental Risk Factors for Unscheduled Hospitalizations of Elderly People
Acronym: RIEHO-C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Virginia BRANCO (Other)
Responsible Party: Sponsor-Investigator, Virginia BRANCO, director of value creation, University of Versailles
Organization: University of Versailles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACE ICSEN 17PIA725
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Environmental Exposure; Individual Difference

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective cohort for etiological and prognostic purposes (Experimental)
  Interventions: Other: Prospective cohort for etiological and prognostic purposes

INTERVENTIONS:
Other: Prospective cohort for etiological and prognostic purposes — Subjects benefit from a standardized, comprehensive geriatric evaluation in accordance with the recommendations of good practice during a geriatric consultation. It is completed by a measurement of the gripping force using a dynamometer and a measurement of the respiratory parameters (vital capacity) using a spirometer. The following acts are added to the consultation: the completion of questionnaires, a semi-directed interview focused on the perception of air pollution, the wearing on the chest for one week of an individual mobile physiological signal sensor (DM with CE marking) and the wearing (on the belt or in a bag) for one week of a portable device with two air pollution sensors.

SUMMARY:
The elderly are weakened by the accumulation of chronic diseases. Their acute decompensation often leads to unscheduled hospitalization, which constitutes a breach of care with often serious consequences in terms of morbidity and mortality. Few studies have identified all the risk factors for unscheduled hospitalization in the very elderly. This project deals with the impact of air pollution on the very elderly as a source of physiological decompensations leading to unscheduled hospitalizations, in association with other individual and environmental risk factors. It complements the Rieho cohort that followed 973 elderly people on the same objective and enriches it with the use of sensors measuring the peri-individual atmospheric environment.

DETAILED DESCRIPTION:
In order to facilitate the perspective and scientific valorization of these data, the experimental design and population characteristics reproduce those of the RIEHO cohort (Coordinator P Aegerter), which aims to identify individual and environmental risk factors for unscheduled hospitalization of the elderly and included 973 people over 80 years of age with a 2-year follow-up, closed in early 2017. Indeed, the workforce mobilized in the Rieho-C study is undersized to measure an association between air quality and a major health impact (hospitalization or death), this objective can only be achieved by adding Rieho-C data to those of Rieho.

ELIGIBILITY:
Inclusion Criteria:

* Person over 80 years of age consulting in the geriatrics department of Ste-Périne Hospital (Gerontology Consultations, Dr A Hiance- Delahaye, Head of Department Pr J Ankri. Paris XVI), for a standardised geriatric assessment, for any reason, if it does not result in immediate or foreseeable hospitalisation within 2 weeks,
* Living at home or in a residence,
* Subject living in Ile-de-France,
* Subject speaking French; this study requires minimal participation of subjects (wearing sensors, qualitative interview) that does not appear compatible with comprehension problems,
* MMSE Score ≥ 15
* ADL score ≥ 3
* Affiliated with a health insurance plan or eligible,
* Person who has signed an informed and written consent.

Exclusion Criteria:

* Subject whose state of health requires hospitalization within two weeks,
* Subject under guardianship or curatorship,
* Subject living in collective housing (retirement home) or entering an institution within 2 weeks,
* Abundant thoracic hair causing poor contact of the ECG electrodes of the physiological sensor,
* Rejection of patient's contact information, refuses to answer questionnaires and follow-up visits, or refuses to wear sensors, Impossibility, during the initial assessment, to establish at least telephone contact with the caregiver when he or she organizes the home visit,
* Subject already included in the study.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
To describe the quality of the peri-individual atmospheric environment, both indoor and outdoor | 3 years
  The quality of the peri-individual atmospheric environment will be described by the distribution (average, maximum and cumulative values) of the daily concentrations of pollutants (PM10, NO2).